CLINICAL TRIAL: NCT03221998
Title: The Effect of Timing of Intravenous Paracetamol Administration on Post-surgical Pain and Cytokines Levels Following Laparoscopic Sleeve Gastrectomy
Brief Title: The Effect of Timing of Intravenous Paracetamol Administration on Post-surgical Pain
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Yair Binyamin MD, principal lnvestigator, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sor17ybyrctil
Record Dates: First submitted 2017-06-30; First posted 2017-07-19 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Obesity, Morbid
Keywords: morbidly obese; ,elective sleeve; gastrectomy; paracetamol; IV Perfelgan
MeSH Terms: conditions — Obesity, Morbid | interventions — Acetaminophen; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: This study is designed as a population-based prospective randomized cohort study. A prospective cohort of patients admitted to laparoscopic sleeve gastrectomy due to morbid obesity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV paracetamol (Experimental): Patients in the first group will receive in the operating room before surgery 1 gram (100 ml) of intravenous paracetamol ( IV paracetamol) for 15 minutes intraoperative
  Interventions: Drug: IV paracetamol
- IV saline (NaCl 0.9 %) (Placebo Comparator): Patients in the second group will receive 100 mL NACL 0.9% (IV NaCl 0.9 %)intraoperative
  Interventions: Drug: IV saline (NaCl 0.9 %)

INTERVENTIONS:
Drug: IV paracetamol — 100 gram paracetamol infusion for moderate pain management
  Other Names: Perfalgan infusion (paracetamol)
  Arms: IV paracetamol
Drug: IV saline (NaCl 0.9 %) — 100 ml of Normal Saline (IV NaCl 0.9 %) as placebo
  Other Names: Normal Saline
  Arms: IV saline (NaCl 0.9 %)

SUMMARY:
This study is designed as a population-based prospective randomized cohort study. A prospective cohort of patients admitted to laparoscopic sleeve gastrectomy due to morbid obesity

DETAILED DESCRIPTION:
All adult consecutive patients admitted to surgical departments for laparoscopic sleeve gastrectomy will be enrolled prospectively.

For the purposes of the current study we want to determine how much paracetamol (acetaminophen) can reduce the cytokines levels in these patients

The study enrollment period is planned to be a year. The follow-up period for each patient will be until discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients admitted for laparoscopic sleeve gastrectomy
* Elective surgery
* BMI > 40
* American Society of Anesthesiology Classification: 1-2

Exclusion Criteria:

* Patients' refusal to participate in the study
* Patients unable to give an informed consent
* Pregnancy
* Emergency surgery
* Patient with known allergy to paracetamol
* Patient with hepatic failure
* international normalized ratio >1.7
* Albumin<3.5g/Dl
* Bilirubin >2mg/dL
* Patient with fever > 37.5 ° C
* Patient with hemoglobin < 8
* Patients chronically treated with steroids or steroid-treated patients over a month in the year preceding surgery.

Drug addict

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
measuring of Visual Analogue pain Scale, | up to 48 hours after surgery
  Visual Analogue pain Scale to determine patient level of pain , for establish the correct timing of paracetamol administration
measuring of Cytokine levels | up to 48 hours after surgery
  measuring of Cytokine levels in comparison of timing of paracetamol administration , as a predictor for inflammatory mediators released in response to noxious stimuli

SECONDARY OUTCOMES:
Total consumption of opiates after surgery | up to 72 hours after surgery
  post - operative opioid consumption in manner of dosage and frequency in ward
Respiratory post-operative complication while in ward | up to 72 hours after surgery
  Respiratory complication (need of respiratory support, need of intensive care unit hospitalization)
septic post-operative complication while in ward | up to 72 hours after surgery
  development of fever above 38° C
Cardiovascular post-operative complication while in ward | up to 72 hours after surgery
  Cardiovascular complication (hemodynamic instability, inotropic support )
Gastrointestinal post-operative complication while in ward | up to 72 hours after surgery
  Gastrointestinal complaints as nausea and vomiting, need to use antiemetic drug
urinary trak post-operative complication while in ward | up to 72 hours after surgery
  Incidence of urinary retention and need for catheterization
post-operative pruritus while in ward | up to 72 hours after surgery
  Pruritus
post-operative hospitalization | up to one week after surgery
  length of hospital stay by number of days
Respiratory post-operative complication while recovering in post anesthesia care unit | up to 5 hours after surgery
  Respiratory complication need of respiratory support, need of intensive care unit hospitalization)
septic post-operative complication while recovering in post anesthesia care unit | up to 5 hours after surgery
  Development of fever above 38° C
Cardiovascular post-operative complication while recovering in post anesthesia care unit | up to 5 hours after surgery
  Cardiovascular complication (hemodynamic instability, inotropic support )
Gastrointestinal post-operative complication while recovering in post anesthesia care unit | up to 5 hours after surgery
  Gastrointestinal complication as nausea and vomiting, need to use antiemetic drugs
urinary retention post-operative complication while recovering in post anesthesia care unit | up to 5 hours after surgery
  incience of urinary retention and need for catheterization
post-operative pruritus while recovering in post anesthesia care unit | up to 5 hours after surgery
  Pruritus
post-operative stay in post anesthesia care unit | up to 5 hours after surgery
  length of post anesthesia care unit stay by number of hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Semionov, MD, Study Director — Soroka University Medical Center-Department of Anesthesiology; Alexander Zlotnic, PhdMD, Study Chair — Soroka University Medical Center-Department of Anesthesiology; Yair Binyamin, MD, Principal Investigator — Soroka University Medical Center-Department of Anesthesiology; Yair Yaish Reina, MD, Principal Investigator — Soroka University Medical Center-Department of Anesthesiology

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ruiz-Tovar J, Munoz JL, Gonzalez J, Zubiaga L, Garcia A, Jimenez M, Ferrigni C, Duran M. Postoperative pain after laparoscopic sleeve gastrectomy: comparison of three analgesic schemes (isolated intravenous analgesia, epidural analgesia associated with intravenous analgesia and port-sites infiltration with bupivacaine associated with intravenous analgesia). Surg Endosc. 2017 Jan;31(1):231-236. doi: 10.1007/s00464-016-4961-3. Epub 2016 May 13. PMID 27177956
- [Result] Salihoglu T, Salihoglu Z, Zengin AK, Taskin M, Colakoglu N, Babazade R. The impacts of super obesity versus morbid obesity on respiratory mechanics and simple hemodynamic parameters during bariatric surgery. Obes Surg. 2013 Mar;23(3):379-83. doi: 10.1007/s11695-012-0783-0. PMID 23054575
- [Result] Rieg AD, Stoppe C, Rossaint R, Coburn M, Hein M, Schalte G. [EzPAP(R) therapy of postoperative hypoxemia in the recovery room : experiences with the new compact system of end-expiratory positive airway pressure]. Anaesthesist. 2012 Oct;61(10):867-74. doi: 10.1007/s00101-012-2083-4. Epub 2012 Sep 27. German. PMID 23011043
- [Result] Cullen A, Ferguson A. Perioperative management of the severely obese patient: a selective pathophysiological review. Can J Anaesth. 2012 Oct;59(10):974-96. doi: 10.1007/s12630-012-9760-2. Epub 2012 Jul 26. PMID 22833138
- [Result] Aubrun F, Mazoit JX, Riou B. Postoperative intravenous morphine titration. Br J Anaesth. 2012 Feb;108(2):193-201. doi: 10.1093/bja/aer458. PMID 22250276
- [Result] Macintyre PE, Loadsman JA, Scott DA. Opioids, ventilation and acute pain management. Anaesth Intensive Care. 2011 Jul;39(4):545-58. doi: 10.1177/0310057X1103900405. PMID 21823370
- [Result] Schug SA, Raymann A. Postoperative pain management of the obese patient. Best Pract Res Clin Anaesthesiol. 2011 Mar;25(1):73-81. doi: 10.1016/j.bpa.2010.12.001. PMID 21516915
- [Result] Daszkiewicz A, Wylezol M. Postoperative analgesia in a morbidly obese patient with chronic renal failure. Anestezjol Intens Ter. 2010 Oct-Dec;42(4):197-200. PMID 21252836
- [Result] Ahmed S, Morrow E, Morton J. Perioperative considerations when operating on the very obese: tricks of the trade. Minerva Chir. 2010 Dec;65(6):667-75. PMID 21224800
- [Result] Pelosi P, Gregoretti C. Perioperative management of obese patients. Best Pract Res Clin Anaesthesiol. 2010 Jun;24(2):211-25. doi: 10.1016/j.bpa.2010.02.001. PMID 20608558
- [Result] Hans GA, Lauwick S, Kaba A, Brichant JF, Joris JL. Postoperative respiratory problems in morbidly obese patients. Acta Anaesthesiol Belg. 2009;60(3):169-75. PMID 19961114
- [Result] Bodian CA, Freedman G, Hossain S, Eisenkraft JB, Beilin Y. The visual analog scale for pain: clinical significance in postoperative patients. Anesthesiology. 2001 Dec;95(6):1356-61. doi: 10.1097/00000542-200112000-00013. PMID 11748392
- [Result] Heinrich S, Horbach T, Salleck D, Birkholz T, Irouschek A, Schmidt J. [Perioperative anaesthesiological management in 167 patients undergoing bariatric surgery]. Zentralbl Chir. 2011 Dec;136(6):604-11. doi: 10.1055/s-0031-1271382. Epub 2011 Apr 14. German. PMID 21495003